CLINICAL TRIAL: NCT02363491
Title: A Prospective, Open Label Phase I/II Study to Assess the Safety and Efficacy of Cycles of Intravenously Infused Doses of OPN-305 in Second-line or Third-line Lower (Low and Intermediate-1) Risk Myelodysplastic Syndrome (MDS)
Brief Title: A Phase I/II Study of OPN-305 in Second-line Lower Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Opsona Therapeutics Ltd. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Montefiore Medical Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN-305-106
Record Dates: First submitted 2015-01-21; First posted 2015-02-16 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — tomaralimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OPN-305 (Experimental): OPN-305
  Interventions: Drug: OPN-305

INTERVENTIONS:
Drug: OPN-305 — For the dose confirming part of the study, patients will receive a starting dose of 5 mg/kg OPN-305.

SUMMARY:
The dose-confirming part of this study, comprising at least 10 patients is designed as a single center, prospective, single arm, open label in patients who have failed or are unresponsive to Azacitidine (AZA) or Decitabine (they may also have additionally failed an Erythropoiesis Stimulating Agent (ESA) followed by a dose expansion part with at least 44 patients; the objective of the whole study being to assess the safety, efficacy, pharmacokinetics and pharmacodynamics of intravenously infused multiple doses of OPN-305 in low and intermediate-1 risk myelodysplastic syndrome (second and third line Lower risk MDS).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Diagnosis of MDS (de novo or secondary) by bone marrow aspirate based on the World Health Organization (WHO) classification - Low and Intermediate-1 risk categories MDS using the IPSS (International Prognostic Scoring System)
* AZA/decitabine (this applies to standard of care and investigational drugs) failure (Dose confirming and Dose expansion parts):
* defined as discontinuation due to any of the following:

  * Lack of response after at least 4 cycles
  * Loss of response (patient must have received therapy for at least 4 cycles)
  * Progressive disease
  * Adverse events

Note: Patients are eligible if additionally they have failed an ESA

* HMA Naïve group:

  * Never received a hypomethylating agent for MDS
  * Failed or ceased to respond to ESA(s)
  * ESA ineligible; defined as endogenous serum erythropoietin level > 200 U/L for subjects not previously treated with ESAs
* Red blood cell transfusion dependent defined as ≥ 2 Red blood cells (RBC) units required in the 8 weeks prior to starting in the study. In addition, there should be no 8 consecutive weeks without red blood cell transfusions in the 16 weeks prior to enrolment.
* Life expectancy ≥ 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status Grade 0-2
* Serum bilirubin levels ≤2 x upper limits of normal (ULN)
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤2.5 x ULN
* Del 5q patients who have failed or are not eligible for Revlimid
* Creatinine clearance >30 ml/min calculated by the Cockcroft-Gault formula
* Willingness to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations
* Negative urine β-human chorionic gonadotropin (β-HCG) pregnancy test for fertile women at screening and confirmed by serum pregnancy test in the 48 hours prior to OPN-305 administration
* If sexually active female, patient must be/have one of the following:
* Post-menopausal defined as the absence of menses for at least one year (serum Follicle-stimulating hormone (FSH) ≥20IU/L can also be measured according to local practice),OR
* Surgically sterile defined as a bilateral tubal ligation at least 6 months prior to administration of study drug, bilateral oophorectomy, or complete hysterectomy, OR
* Using an effective means of contraception that is planned to continue for the duration of treatment and for a further 3 months.
* If sexually active male, patient must: Agree to use an effective means of contraception (per site-specific guidelines) that is planned to continue until 6 months after the last dose of OPN-305.Agree not to donate sperm until 6 months after the last dose of OPN-305

Exclusion Criteria:

* Diagnosis of MDS by bone marrow aspirate of Intermediate-2 and High risk category MDS based on the World Health Organization (WHO) classification using the IPSS (International Prognostic Scoring System)
* Patients with 5q deletion (del) MDS eligible for Revlimid (lenalidomide)
* Hypomethylating agent (HMA) Naïve group:

  * Have received a hypomethylating agent for MDS
  * Have not failed or ceased to respond to an ESA
  * Are not ESA ineligible as defined in inclusion criteria
* Prior history of acute leukemia or AML
* Unable/unwilling to undergo bone marrow sampling
* Prior history of bone marrow transplantation
* Prior malignancy (other than non-invasive malignancy including in situ cervical cancer, Bowen's disease, basal cell cancer of the skin and non-invasive or excised skin squamous cell carcinoma) unless treated with curative intent and without evidence of disease for 3 years before randomization
* Active viral or bacterial infections: this includes any infections that are being actively treated even if the signs and symptoms appear to have resolved. Courses of antibiotics or anti-viral treatment should be completed before the patients is enrolled
* Unstable angina, congestive heart failure [NYHA (New York Heart Association) >class II], uncontrolled hypertension [diastolic > 100 mmHg], uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction, uncontrolled diabetes mellitus
* Clinical Evidence of Central Nervous System (CNS) disease
* Less than 4 weeks since any therapy for MDS
* Prior history of anaphylaxis to similar products
* History or presence of a medical condition or disease or substance abuse that in the investigator's assessment would place the patient at an unacceptable risk for study participation
* Lactating or pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Establishment of the dose and dose frequency based on dose-limiting toxicity and bone marrow receptor occupancy of OPN-305 in low and intermediate -1 (Lower) risk MDS | 8 weeks
Tolerability of OPN-305 as monotherapy based on adverse events | 16 weeks/32 weeks (if there is no AZA add-back)
Tolerability of OPN-305 as monotherapy and in combination with AZA based on adverse events | 32 weeks

SECONDARY OUTCOMES:
Hematological response based on International Working Group (IWG) 2000/2006 | week 36
Cytokine levels in serum (TNFα, IL-1β, IL-6, IL-10, IL-12, IL-18, IL-23 and IFN-γ) | day 1 and week 4
Immunogenicity of OPN-305 (Measurement of anti drug antibodies and neutralizing antibodies) | day 1, weeks 4, 8, 16, 24 and 32
Incidence of infections | 36 weeks
Pharmacokinetic profile of OPN-305 (maximum concentration (Cmax)) | day 1, weeks 4, 8, 12, 16, 20, 24, 28, 32
Pharmacokinetic profile of OPN-305 (time at which Cmax is attained (tmax)) | day 1, weeks 4, 8, 12, 16, 20, 24, 28, 32
OPN-305 receptor occupancy in peripheral monocytes, bone marrow cells and stroma | screening (bone marrow only), day 1 (blood only), wks 4 (blood only), 8, 12 (blood only), 16, 20 (blood only), 24 (blood only), 28 (blood only), 32 and 36 (blood only)
Correlation of clinical response with cytogenical observations | wk 36
Quality of life MD Anderson Symptom Inventory (MDASI) - Acute Myeloid Leukemia (AML)/Myelodysplastic syndrome (MDS) questionnaire | wk 36
  MDASI is MD Anderson symptom inventory. It has two scales
  1. Severity of symptoms scale 0-10 with 0 being not present and 10 being as bad as you can imagine
  2. How symptoms interfere with life scale 0-10 with 0 did not interfere and 10 interfere completely

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Research Site, Tampa, Florida
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Houston, Texas